CLINICAL TRIAL: NCT07320105
Title: Efficacy of Postoperative Radiotherapy in Patients With Multiple Postoperative N2 Metastases From Non-Small Cell Lung Cancer in the Immunotherapy Era: A Multicenter Prospective Controlled Phase II Clinical Trial
Brief Title: Postoperative Radiotherapy for Postoperative N2 Metastases of NSCLC in the Immunotherapy Era (Phase II)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-RT-2025
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + Chemotherapy Arm (Experimental): This arm includes postoperative non-small cell lung cancer patients receiving Tislelizumab (standard intravenous dose) combined with platinum-based chemotherapy (adjuvant regimen), without additional radiotherapy.
  Interventions: Drug: Tislelizumab + platinum-based chemotherapy
- Tislelizumab + Chemotherapy + Radiotherapy Arm (Experimental): This arm includes postoperative non-small cell lung cancer patients receiving Tislelizumab + platinum-based chemotherapy (same as Group A), plus focal radiotherapy (50Gy to the lesion area).
  Interventions: Drug: Tislelizumab + platinum-based chemotherapy + focal radiotherapy

INTERVENTIONS:
Drug: Tislelizumab + platinum-based chemotherapy — Tislelizumab (200mg IV every 3 weeks) combined with platinum-based chemotherapy (postoperative adjuvant regimen).
  Arms: Tislelizumab + Chemotherapy Arm
Drug: Tislelizumab + platinum-based chemotherapy + focal radiotherapy — Tislelizumab + platinum-based chemotherapy (same as above) plus focal radiotherapy (50Gy total dose to the lesion).
  Arms: Tislelizumab + Chemotherapy + Radiotherapy Arm

SUMMARY:
This study will be conducted at Fujian Provincial Cancer Hospital. Its main goals are to evaluate the progression-free survival (PFS) and safety of postoperative immunotherapy combined with radiotherapy in patients with high-risk stage Ⅲ N2 non-small cell lung cancer after surgery. It will also assess the overall survival (OS) of this treatment as a secondary goal.

This study has been approved by the Medical Ethics Committee of Fujian Provincial Cancer Hospital, and the rights and safety of all participants will be fully protected during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old and ≤75 years old, no gender restriction; Pathologically (histologically or cytologically) confirmed non-small cell lung cancer with multiple N2 metastasis after surgery; No prior radiotherapy, chemotherapy or immunotherapy; At least 3 lymph node metastases confirmed by postoperative pathology; ECOG PS score: 0-2; Expected survival time ≥3 months; Normal major organ function, with basically normal results of blood routine, blood biochemistry and coagulation function tests; Basically normal immune indicators; No severe underlying diseases or severe cardiopulmonary dysfunction.

Exclusion Criteria:

* Known or suspected active autoimmune diseases, or history of autoimmune diseases (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, etc.); History of immunodeficiency (including positive HIV test), other acquired/congenital immunodeficiency diseases, organ transplantation or allogeneic bone marrow transplantation; Interstitial lung disease, drug-induced pneumonia, radiation pneumonia requiring steroid treatment, symptomatic active pneumonia, or severe pulmonary dysfunction; Poorly controlled cardiovascular symptoms or diseases (e.g., NYHA class II or higher heart failure, unstable angina, myocardial infarction within 1 year, uncontrolled arrhythmia); Active hepatitis B (HBV DNA ≥2000 IU/mL or 10⁴ copies/mL) or hepatitis C (positive anti-HCV and HCV-RNA above detection limit); Hereditary bleeding tendency or coagulation dysfunction; bleeding symptoms within 3 months, or positive fecal occult blood (++ or above); Toxicity from prior anti-tumor therapy not recovered to ≤CTCAE grade 1 (except alopecia); Known or suspected allergy to the study drug; Pregnant or lactating women; Subjects deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Every 3 months, up to 24 months after randomization
  The time from randomization to the first occurrence of disease progression (per RECIST 1.1 criteria) or death from any cause; assessed every 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
At the current stage, the IPD sharing plan has not yet been finalized. Following study completion, we will conduct a comprehensive evaluation of data sharing feasibility-including considerations related to participant privacy protection, data standardization, and regulatory compliance-before determining a specific sharing framework based on study progress and relevant requirements.